CLINICAL TRIAL: NCT04360421
Title: Use of Liposomal Bupivacaine (Exparel) In Expedited Recovery Following Lower Extremity Amputation
Brief Title: Use of Long-acting Bupivacaine In Lower Extremity Amputation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5200004
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Amputation; Anesthesia, Local; Opioid Use
Keywords: lower extremity amputation; liposomal bupivacaine; expedited recovery; vascular surgery; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intraoperative liposomal bupivacaine field block (Experimental): Patients will receive the maximum dosage of liposomal bupivacaine allowed for their body weight or the full vial, whichever is less. Injected once, along the incision before closure of the skin.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Patient's undergoing major extremity amputation and enrolled in the study as part of the experimental arm will, during their amputation operation, receive liposomal bupivicaine per recommended manufacturing dosing and administration in a "field block" for long-acting local anesthesia.

SUMMARY:
The purpose of this investigator-initiated study is to assess the use of liposomal bupivacaine in major extremity amputation and its effects on post-operative opioid narcotic use, length of stay, and in-hospital costs. Liposomal bupivacaine is an encapsulated, injectable amide anesthetic intended for use in long-acting local anesthesia. It has been shown in randomized trials to be effective in reducing post-operative pain while reducing opioid narcotic use and length of hospital stay following several surgical procedures, particularly after total knee arthroplasty. Extremity amputation is a painful operation often performed in seriously ill or debilitated patients, often related to infection, trauma or malignancy. Application of liposomal bupivacaine in extremity amputation is not well described. The investigators intend to enroll adults greater than age 18 years of age who are to undergo major extremity amputation. Patients will receive targeted injections of liposomal bupivacaine during their procedure. Patient pain scores, total opioid use, and length of hospital stay will be tracked. Patients receiving liposomal bupivicaine will be compared to similarly matched subjects who received standard anesthesia regimens without liposomal bupivicaine. The investigators hypothesize that liposomal bupivicaine used during major amputation decreases opioid use, hospital stay, and in-hospital costs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients who underwent unilateral or bilateral lower extremity major amputation, either primary or revision: partial foot, ankle disarticulation, transtibial, knee disarticulation, transfemoral [1 year retrospective analysis]
* Patients who meet clinical indication for unilateral or bilateral lower extremity major amputation, either primary or revision: partial foot, ankle disarticulation, transtibial, knee disarticulation, transfemoral

Exclusion Criteria:

* Minor amputations
* Liver dysfunction (impaired metabolism of Amides)
* Concomitant psychiatric or chronic pain disorders
* Pregnancy
* Amide anesthetic allergy
* Presence of perioperative sepsis or acute organ dysfunction
* Need for ICU admission at any point
* Polytrauma
* Quadriplegic/Paraplegic/Insensate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Total opioid use | Up to 4 weeks
  Total morphine equivalent
Total cost of stay | Up to 4 weeks
  US Dollar cost

SECONDARY OUTCOMES:
Pain scores | Up to 4 weeks
  Numeric rating scale of 0 to 10, where 0 is no pain and 10 is the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kristyn Mannoia, MD, Principal Investigator — Loma Linda University Department of Vascular Surgery
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motakef S, Wong WW, Ingargiola MJ, Nguyen D, Galdyn IA, Kim HY, Gupta SC. Liposomal Bupivacaine in Implant-Based Breast Reconstruction. Plast Reconstr Surg Glob Open. 2017 Nov 20;5(11):e1559. doi: 10.1097/GOX.0000000000001559. eCollection 2017 Nov. PMID 29263963
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Background] Hyland SJ, Deliberato DG, Fada RA, Romanelli MJ, Collins CL, Wasielewski RC. Liposomal Bupivacaine Versus Standard Periarticular Injection in Total Knee Arthroplasty With Regional Anesthesia: A Prospective Randomized Controlled Trial. J Arthroplasty. 2019 Mar;34(3):488-494. doi: 10.1016/j.arth.2018.11.026. Epub 2018 Nov 23. PMID 30554925
- [Background] Felling DR, Jackson MW, Ferraro J, Battaglia MA, Albright JJ, Wu J, Genord CK, Brockhaus KK, Bhave RA, McClure AM, Shanker BA, Cleary RK. Liposomal Bupivacaine Transversus Abdominis Plane Block Versus Epidural Analgesia in a Colon and Rectal Surgery Enhanced Recovery Pathway: A Randomized Clinical Trial. Dis Colon Rectum. 2018 Oct;61(10):1196-1204. doi: 10.1097/DCR.0000000000001211. PMID 30192328
- [Background] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785